CLINICAL TRIAL: NCT05500547
Title: Clinical Performance of One-shade Universal Dental Resin Composite as Posterior Restoration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ruba Salah Anwar, Assistant Lecturer at Department of Operative Dentistry, Faculty of Dentistry, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RSAnwar
Record Dates: First submitted 2022-07-26; First posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Carious Teeth
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Universal single shade resin composite restorative material (Experimental): Dental restorative material
  Interventions: Other: US Public Health Service "USPSH" criteria for assessment of success of resin composite restorations
- Nano-hybrid multi-shade resin composite restorative material (Active Comparator): Dental restorative material
  Interventions: Other: US Public Health Service "USPSH" criteria for assessment of success of resin composite restorations

INTERVENTIONS:
Other: US Public Health Service "USPSH" criteria for assessment of success of resin composite restorations — US Public Health Service "USPSH" criteria for color match, marginal adaptation, surface texture, retention, recurrent caries and others after 1, 3, 6 and 9 months.
  Other Names: assessment of Universal single shade resin composite and Nano-hybrid multi-shade resin composite restorative material using the US Public Health Service "USPSH" criteria

SUMMARY:
This study is aimed to evaluate the clinical performance of new One-shade universal composite resin as posterior restoration using US Public Health Service "USPSH" criteria for color match, marginal adaptation, surface texture, retention, recurrent caries and others after 1, 3, 6 and 9 months.

DETAILED DESCRIPTION:
One operator will place all restorations under rubber-dam isolation. The patients will receive restorations with both materials, randomly after shade selection (The shade of single shade universal resin composite "Omnichroma" will be taken before and after placement into the cavity). During the referred period, only the two composites in study will be placed in posterior teeth in the dental office. The various materials' application procedure will be applied according to manufacturer's instructions.

ELIGIBILITY:
Inclusion Criteria:

* • They should have an acceptable oral hygiene level.

  * Presence of at least two occlusal carious lesions to be restored with two different types of composite.
  * The two studied materials restorations should be used in approximately the same sized lesions or within the same extension.
  * Age range between 25 and 45years.

Exclusion Criteria:

* • Severe or active periodontal or carious disease and heavy bruxism or a traumatic occlusion

  * Patients with a compromised medical history, or had received therapeutic irradiation to the head and neck region.
  * Alcoholic and smoker patients.
  * Patients had participated in a clinical trial within 6 months before commencement of this trial.
  * Patients unable to return for recall appointment

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
USPSH criteria | For 9 months
  Alpha and Beta are clinically successful, Charlie and Delta are clinically failure

CONTACTS AND LOCATIONS:
Overall Officials: Mona I Riad, Prof, Study Director — Minia University
Locations (1):
- Ruba Salah Anwar, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol